CLINICAL TRIAL: NCT00292474
Title: TAXUS IV-SR: Treatment of De Novo Coronary Disease Using a Single Paclitaxel-Eluting Stent
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Kristan Tilton, Boston Scientific
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2004; TAXUS IV
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary interventions; stent implant; drug-coated stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- TAXUS Express (Experimental)
  Interventions: Device: percutaneous coronary intervention
- Express Bare (Placebo Comparator)
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention

SUMMARY:
The ultimate goal of a paclitaxel eluting stent system (TAXUS stent) is to prevent restenosis by blunting the initial response to stent implant injury and sustaining the arrested response until vascular healing has taken place.

The purpose of the TAXUS IV-SR trial is to study the safety and efficacy of the TAXUS Stent under controlled trial circumstances used in the treatment of new coronary artery lesions (heart blockages) This clinical investigation will evaluate the safety and effectiveness of the TAXUS Stent with 1 ug/mm2 (loaded drug/stent surface area) of paclitaxel incorporated into a slow rate-release formulation of a triblock copolymer carrier system for treatment of new coronary artery lesions.

DETAILED DESCRIPTION:
This was a prospective randomized, double-blind, multicenter safety and efficacy trial. Patients were stratified by presence or absence of medically treated diabetes mellitus and vessel diameter (<3.0 mm or >/=3.0 mm), then randomized 1:1 to receive either the TAXUS Stent or a Control stent. Additional study stents were permitted to optimize outcomes. The study was considered complete (with regard to the primary endpoint) after all patients enrolled had completed the 9 month follow-up.

Enrollment of 1172 patients was planned; 1326 were treated and randomized at 73 centers involving 76 sites by 8 July 2002 with 667 in the TAXUS group and 659 in the Control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > or = 18 years old
2. Eligible for percutaneous coronary intervention (PCI)
3. Documented stable angina pectoris (Canadian Cardiovascular Society Classification [CCS] 1, 2, 3, or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
4. Left ventricular ejection fraction (LVEF) of > or = 25%
5. Acceptable candidate for CABG
6. Patient (or legal guardian) understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
7. Willing to comply with all specified follow-up evaluations

1. Target lesion located within a single native coronary vessel 2. Target lesion randomized to treatment with the study device may be composed of multiple lesions but must be completely coverable by one (1) study stent 3. Cumulative target lesion length is > or = 10 mm and < or = 28 mm (visual estimate) 4. RVD of > or = 2.5mm to < or = 3.75 mm (visual estimate) 5. Target lesion diameter stenosis > or = 50% (visual estimate) 6. Target lesion is de novo (i.e., a coronary lesion not previously treated)

7. Target lesion located within a single native coronary vessel 8. Target lesion randomized to treatment with the study device may be composed of multiple lesions but must be completely coverable by one (1) study stent 9. Cumulative target lesion length is > or = 10 mm and < or = 28 mm (visual estimate) 10. RVD of > or = 2.5mm to < or = 3.75 mm (visual estimate) 11. Target lesion diameter stenosis > or = 50% (visual estimate) 12. Target lesion is de novo (i.e., a coronary lesion not previously treated)

-

Exclusion Criteria:

1. Known sensitivity to paclitaxel 2. Any previous or planned treatment with a non-study anti-restenotic drug-coated or drug-eluting coronary stent. (Note: previous or planned treatment with heparin or phosphorylcholine coated stents is acceptable, as long as the procedure with the non-study stent meets the protocol defined criteria for staged procedures) 3. Previous or planned treatment with intravascular brachytherapy in the target vessel 4. MI within 72 hours prior to the index procedure and/or CK-MB >2x the local laboratory's upper limits of normal (refers to a measured value on the day of the index procedure) 5. Cerebrovascular Accident (CVA) within the past 6 months 6. Acute or chronic renal dysfunction (creatinine >2.0 mg/dl or >150 µmol/L) 7. Contraindication to ASA, or to both clopidogrel and ticlopidine 8. Leukopenia (leukocyte count <3.5 x 109/liter) 9. Thrombocytopenia (platelet count <100,000/mm3) 10. Active peptic ulcer or active gastrointestinal (GI) bleeding 11. Known allergy to stainless steel 12. Any prior true anaphylactic reaction to contrast agents 13. Known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure 14. Patient is currently taking colchicine 15. Patient is currently, or has been treated with paclitaxel within 12 months of the index procedure 16. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the study 17. Life expectancy of less than 24 months due to other medical conditions 18. Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study 19. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1326 (Actual)
Dates: Start 2002-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety and effectiveness of the TAXUS Stent System with 1 ug/mm2 (loaded drug/stent surface area) of paclitaxel incorporated into a slow rate-release formulation of a triblock copolymer carrier syst

SECONDARY OUTCOMES:
Secondary endpoints include the following:
• Rates of composite MACE and the individual components of MACE (MI, TVR, Cardiac Death), assessed at 1, 4 and 9 months after the index procedure and annually for 5 more years (i.e., 1, 2, 3, 4, and 5 years after the index procedure).
• Stent thrombosis rate
• Target Vessel Failure
• Clinical procedural success
• Binary restenosis rate

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — Columbia Hospital; Stephen G Ellis, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Stephen G.Ellis, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Wakabayashi K, Mintz GS, Weissman NJ, Stone GW, Ellis SG, Grube E, Ormiston JA, Turco MA, Pakala R, Xue Z, Desale S, Laynez-Carnicero A, Romaguera R, Sardi G, Pichard AD, Waksman R. Impact of drug-eluting stents on distal vessels. Circ Cardiovasc Interv. 2012 Apr;5(2):211-9. doi: 10.1161/CIRCINTERVENTIONS.111.965780. Epub 2012 Apr 10. PMID 22496083
- [Derived] Ellis SG, Stone GW, Cox DA, Hermiller J, O'Shaughnessy C, Mann T, Turco M, Caputo R, Bergin PJ, Bowman TS, Baim DS; TAXUS IV Investigators. Long-term safety and efficacy with paclitaxel-eluting stents: 5-year final results of the TAXUS IV clinical trial (TAXUS IV-SR: Treatment of De Novo Coronary Disease Using a Single Paclitaxel-Eluting Stent). JACC Cardiovasc Interv. 2009 Dec;2(12):1248-59. doi: 10.1016/j.jcin.2009.10.003. PMID 20129552